CLINICAL TRIAL: NCT03153852
Title: The Efficacy of Combined Peels in Treatment of Melasma Using Modified Jessner's Solution With 20%Trichloroacetic Acid Versus 70%Glycolic Acid With 20% Trichloroacetic Acid : A Split-face Study
Brief Title: Modified Jessner's Solution With Trichloroacetic Acid Versus Glycolic Acid With Trichloroacetic Acid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereny Ramsis, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: combined peels
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — glycolic acid; Trichloroacetic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined peeling agents (Experimental): Modified Jessner's solution will be applied on the right side and glycolic acid 70% on the other side of the face.trichloroacetic acid 20% will be applied in one uniform coat to both sides
  Interventions: Drug: Modified Jessner's solution; Drug: Glycolic acid; Drug: Trichloroacetic acid

INTERVENTIONS:
Drug: Modified Jessner's solution — Modified Jessner's solution will be applied on the right side until frosting
  Other Names: Combined peel
Drug: Glycolic acid — Glycolic acid 70% on the other side of the face, then it will be neutralized with water after 5 minutes
  Other Names: Combined peel
Drug: Trichloroacetic acid — Trichloroacetic acid 20% will be applied in one uniform coat to both sides of the face until frosting
  Other Names: Combined peel

SUMMARY:
Melasma is a common acquired disorder of hyperpigmentation characterized by irregular light brown to dark brown patches of hyperpigmentation commonly affecting the face. The trunk and arms are also occasionally involved .

DETAILED DESCRIPTION:
Key etiologic factors include a genetic predisposition, solar damage, barrier abnormalities, and unique sensitivities to hormonal changes including pregnancy, oral contraceptives, and hormone replacement therapy .Melasma can be divided into centrofacial, malar, and mandibular, according to the pigment distribution on the skin. The hyperpigmented patches are usually symmetrical and have a sharp irregular border.On wood's light examination three forms of melasma exist (epidermal, dermal, and mixed). Epidermal & mixed types shows accentuation of pigmentation, while there is no change in dermal type The epidermal type is the most responsive to treatment .Melasma is often difficult to treat, and the condition may be refractory. Principles of therapy include protection from ultraviolet light, inhibition of melanocyte activity and melanin synthesis, and the disruption and removal of melanin granules .Many depigmenting agents and other therapies such as chemical peeling are used for treating melasma, in the form of monotherapy or combined therapy .The most commonly used peeling agents are alpha-hydroxy-acids, glycolic acid , Jessner solution, salicylic acid resorcinol,trichloroacetic acid , pyruvic acid and phenol Several hypopigmenting agents such as topical hydroquinone (2 to 4%) alone or in combination with tretinoin (0.05 to 0.1%) have been used with differing results. Topical azelaic acid (15 to 20%) can be as efficacious as hydroquinone. Kojic acid, alone or in combination with glycolic acid or hydroquinone, has shown good results, due to its inhibitory action on tyrosinase. Chemical peeling is apromising treatment for numerous pigmentary disorders as melasma.Which aim to remove the melanin ,rather than the inhibition of melanocytes or melanogenesis by causing controlled necrosis and subsequent regeneration of the epidermis ,apart from remodeling of collagen and elastic fiberes in the dermis . The gold standard for chemical peeling agents is trichloroacetic acid It is a traditional chemical substance which has been used for both superficial and medium-depth as well as deep peelings.It is not expensive, stable, not light-sensitive and does not need to be neutralized .Classic Jessner's solution is a combination of different chemical substances, including salicylic acid(14gm), resorcinol(14gm), lactic acid(14gm) and ethanol, which can be used either alone for superficial peeling or in combination with other agents to make easier medium-depth procedures. Dr.Max Jessner originally formulated this peel to reduce the concentration and toxicity of each of the individual ingredients while increasing efficacy. Modified formula: lactic acid(17%), salicylic acid(17%), citric acid(8%) and ethanol .It is preferred , to avoid possible allergic reactions and hyperpigmentation problems, which may be created by resorcinol, especially in skin types V and VI.Gary Monheit has popularized the combination peel using the classic Jessner's solution combined with trichloroacetic acid , to achieve a more uniform penetration and an excellent peel with a low, safe concentration of trichloroacetic acid Glycolic acid it is one of the most frequently used superficial peeling agent.

It is stable , not light sensitive, inexpensive and easy to administer. Generally it is safe; scarring uncommon; persistent erythema and postpeel hyperpigmentation rarely seen.The depth of a Glycolic acid peel is a function of the concentration,volume and duration of application.Glycolic acid has been used in combination with trichloroacetic acid peels .70% glycolic acid is applied to the skin for 2 minutes.This is then neutralized,followed by the application of 35% trichloroacetic acid peels without any prior acetone scrub.This combination is thought to produce greater neoelastogenesis and less inflammation than Jessner/trichloroacetic acid combination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years old.
2. Clinical diagnosis of melasma.
3. Mental capacity to give informed consent.

Exclusion Criteria:

1. Pregnant females and females on oral contraceptive pills.
2. Patients with a history of hypertrophic scars or keloids.
3. Patients with recurrent herpes infection.
4. Patients with unrealistic expectation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Melasma Area and Severity Index (MASI) | The mean change from the baseline to week-12
  MASI = .3A(D+H) [forhead] + .3A(D+H)[right malar] + .3A(D+H)[left malar] + .1A(D+H)[chin]; A = area, D = darkness, and H = homogeneity. Area is based on percentage of the region covered by melasma using a 1-6 scale. Darkness is determined on a 0-3 scale. Homogeneity is based on a 0-4 scale.

SECONDARY OUTCOMES:
Evaluation of Photographs | change from the baseline to week-12
  Photos were evaluated using the grading of worse, no improvement, mild improvement or marked improvement comparing week 12 to baseline.
Global satisfaction score | change from the baseline to week-12
  by Quartile rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Ereny Ramsis, Master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yalamanchili R, Shastry V, Betkerur J. Clinico-epidemiological Study and Quality of Life Assessment in Melasma. Indian J Dermatol. 2015 Sep-Oct;60(5):519. doi: 10.4103/0019-5154.164415. PMID 26538717
- [Background] Perez MI. The stepwise approach to the treatment of melasma. Cutis. 2005 Apr;75(4):217-22. PMID 15916218
- [Background] Javaheri SM, Handa S, Kaur I, Kumar B. Safety and efficacy of glycolic acid facial peel in Indian women with melasma. Int J Dermatol. 2001 May;40(5):354-7. doi: 10.1046/j.1365-4362.2001.01149.x. PMID 11555002
- [Background] Molinar VE, Taylor SC, Pandya AG. What's new in objective assessment and treatment of facial hyperpigmentation? Dermatol Clin. 2014 Apr;32(2):123-35. doi: 10.1016/j.det.2013.12.008. PMID 24679999
- [Background] Gupta AK, Gover MD, Nouri K, Taylor S. The treatment of melasma: a review of clinical trials. J Am Acad Dermatol. 2006 Dec;55(6):1048-65. doi: 10.1016/j.jaad.2006.02.009. Epub 2006 Sep 28. PMID 17097400
- [Background] Rendon M, Berneburg M, Arellano I, Picardo M. Treatment of melasma. J Am Acad Dermatol. 2006 May;54(5 Suppl 2):S272-81. doi: 10.1016/j.jaad.2005.12.039. PMID 16631968
- [Background] Clark E, Scerri L. Superficial and medium-depth chemical peels. Clin Dermatol. 2008 Mar-Apr;26(2):209-18. doi: 10.1016/j.clindermatol.2007.09.015. PMID 18472062
- [Background] Perez-Bernal A, Munoz-Perez MA, Camacho F. Management of facial hyperpigmentation. Am J Clin Dermatol. 2000 Sep-Oct;1(5):261-8. doi: 10.2165/00128071-200001050-00001. PMID 11702317
- [Background] Landau M. Chemical peels. Clin Dermatol. 2008 Mar-Apr;26(2):200-8. doi: 10.1016/j.clindermatol.2007.09.012. PMID 18472061
- [Background] Khunger N; IADVL Task Force. Standard guidelines of care for chemical peels. Indian J Dermatol Venereol Leprol. 2008 Jan;74 Suppl:S5-12. PMID 18688104
- [Background] Monheit GD. The Jessner's + TCA peel: a medium-depth chemical peel. J Dermatol Surg Oncol. 1989 Sep;15(9):945-50. doi: 10.1111/j.1524-4725.1989.tb03181.x. PMID 2778184
- [Background] Monheit GD. Chemical peels. Skin Therapy Lett. 2004 Feb;9(2):6-11. PMID 14749844
- [Background] Soliman MM, Ramadan SA, Bassiouny DA, Abdelmalek M. Combined trichloroacetic acid peel and topical ascorbic acid versus trichloroacetic acid peel alone in the treatment of melasma: a comparative study. J Cosmet Dermatol. 2007 Jun;6(2):89-94. doi: 10.1111/j.1473-2165.2007.00302.x. PMID 17524124
- [Background] Grimes PE. Melasma. Etiologic and therapeutic considerations. Arch Dermatol. 1995 Dec;131(12):1453-7. doi: 10.1001/archderm.131.12.1453. PMID 7492140